CLINICAL TRIAL: NCT06110325
Title: The Effectiveness of a Cawthorne and Cooksey Exercise Program on Balance, Fear of Falling and Dizziness on Daily Life in Older Adults: A Randomized Controlled Trial
Brief Title: Effects of the Cawthorne and Cooksey Exercise Program on Balance, Fear of Falling and Dizziness on Daily Life in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras PT, PhD, Principal Investigator, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-04/2023
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Older Adults; Accidental Falls; Prevention; Exercise
Keywords: Cawthorne and Cooksey Exercise; Balance; Likelihood of Fall; dizziness; physiotherapy
MeSH Terms: conditions — Motor Activity; Dizziness

STUDY DESIGN:
Intervention Model Description: A one-month assessor-blind randomized controlled trial will be conducted involving 30 seniors with balance deficits. Participants will be divided equally into two groups (intervention and control), each comprising 15 individuals. The intervention group will receive a Cawthorne and Cooksey-based exercise program, while the control group will receive counseling on fall prevention and guidance for maintaining an active and healthy lifestyle through informational leaflets.
Who Masked: Outcomes Assessor
Masking Description: Assessor-blind randomized control trial. A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cawthorne and Cooksey exercise program (Experimental): The exercise program will span one month and will center on the Cawthorne and Cooksey exercises targeting the vestibular system. Each session will be conducted individually and last for twenty minutes. The program will take place three times a week, with the initial session held in person and the subsequent two via video assistance from their homes
  Interventions: Other: Cawthorne and Cooksey exercise program
- Control group (Active Comparator): Information/Education on Fall Prevention and Promoting an Active, Healthy Lifestyle through Informational Leaflets.
  Interventions: Other: Control

INTERVENTIONS:
Other: Cawthorne and Cooksey exercise program — Participants in this group will receive an exercise program based on Cawthorne and Cooksey exercises. The intervention will last for 4 weeks, taking place three times a week, with the first session conducted in person and the remaining two assisted via video from their homes.
  Arms: Cawthorne and Cooksey exercise program
Other: Control — Control group will receive counseling focused on fall prevention and promotion of an active, healthy lifestyle through informational leaflets.
  Arms: Control group

SUMMARY:
Background: The vestibular system plays a crucial role in maintaining balance. Deficiencies in this system can result in instability and an increased risk of falls in older adults, posing a significant global health concern due to associated injuries. The Cawthorne and Cooksey program has demonstrated effectiveness in enhancing balance and reducing falls. This study aims to investigate the program's impact on balance, fear of falling, and dizziness in individuals aged 65 and older. Thirty-two older adults will be assigned to intervention and control groups. The intervention group will undergo a video-supported Cawthorne and Cooksey-based therapy, while the control group will receive counseling on fall prevention and healthy living through leaflets. The 4-week intervention will take place three times a week, including one face-to-face session and one via video. Pre- and post-assessments, along with a one-month follow-up, will be conducted.

DETAILED DESCRIPTION:
Background: The vestibular system is a primary contributor to balance maintenance, serving as the absolute reference point in relation to other structures, including the visual system, labyrinth, and proprioceptive receptors. Any deficiency in these systems is automatically associated with balance disturbances, potentially leading to feelings of instability and an increased risk of falling. Falls among the elderly represent a global health concern due to their association with severe injuries and chronic disability. Annually, around 30% of community-dwelling seniors experience at least one fall, with 10%-20% falling two or more times. Any fall can result in injury, prolonged immobilization, decreased functional capacity, negative psychological impact, and in some cases, even mortality. The Cawthorne and Cooksey exercise program has demonstrated effectiveness in improving balance, reducing falls, and enhancing quality of life.

Aim: This study aims to investigate the effectiveness of Cawthorne and Cooksey exercises in enhancing balance, diminishing the fear of falls, and reducing dizziness in individuals over the age of 65.

Methods/Design: Thirty-two older adults are anticipated to participate in this study. Participants will be divided into two groups (intervention and control). The intervention group will receive therapy based on Cawthorne and Cooksey exercises, while the control group will receive counseling focused on fall prevention and promotion of an active, healthy lifestyle through informational leaflets. The intervention will span 4 weeks, occurring three times a week, with the first session conducted in person and the remaining two via video assistance from their homes. Participants' balance, fear of falling, and dizziness will be assessed both before and after the intervention, and re-evaluated one-month post-intervention.

Expected results: This exercise program is expected to significantly benefit elderly individuals by improving their balance and reducing the fear of falling within this specific age group. Additionally, we hypothesize that these exercises will alleviate dizziness and enhance overall quality of life, as supported by existing literature.

ELIGIBILITY:
Inclusion Criteria

* Minimum age of 65 years
* Individuals with a Berg Balance Scale score less than 45
* Persistent dizziness for at least one month
* Individuals who have provided written consent for their participation

Exclusion Criteria:

* Individuals with dementia
* Individuals with cancer
* Individuals with multiple cardiovascular diseases
* Individuals unable to move independently even with the use of an aid.
* Individuals diagnosed with a neurodegenerative disease (e.g., Parkinson's disease)
* Individuals who have recently experienced a stroke
* Recent surgery
* Epilepsy
* History of psychiatric disorders

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in balance will be assessed using the Berg Balance Scale (BBS) | pre-intervention, 4th week, 1-month follow-up
  The BBS, proposed by Berg (Berg et al., 1989; Berg et al., 1992), assesses balance in the elderly. It comprises 14 tests of increasing difficulty, requiring subjects to hold positions or perform specific tasks. Each test is graded from 0 to 4 points, reflecting the examinee's balancing ability (0 indicates low, while 4 indicates high ability). According to Berg et al. (1992), a score of 56 indicates functional balance, while a score below 45 signifies significant balance deficits associated with an increased fall risk. Studies demonstrate strong intra-rater and inter-rater reliability in elderly populations, with intraclass correlation (ICC) ranging from .98 to .88 (Berg et al. 1992), and high content validity (Telenius et al., 2015).
Changes in the fear of falling will be assessed using the Falls Efficacy Scale International (FES-I) | pre-intervention, 4th week, 1-month follow-up
  The FES-I is a validated measure of concerns about falling, designed for use in both research and clinical settings. This questionnaire comprises 16 items and is particularly suitable for research as well as for clinical practice. Scores on the scale range from a minimum of 16 (indicating minimal concern about falling) to a maximum of 64 (indicating pronounced apprehension about falling), with higher scores indicating an elevated fear of falling. In this study, we will utilize the Greek version of the questionnaire, as validated by Billis et al. (2011).
Changes in the impact of dizziness on daily life will be assessed using The Dizziness Handicap Inventory questionnaire (DHI). | pre-intervention, 4th week, 1-month follow-up
  The DHI, questionnaire comprises 25 questions aimed at swiftly gauging the influence of dizziness. These questions are categorized into three sections representing functional, emotional, and physical aspects of dizziness and unsteadiness. Respondents can choose from three options: "Always" (worth 4 points), "Sometimes" (worth 2 points), or "No" (worth 0 points). Following completion, the scores for each question are totaled, resulting in a score ranging from 0 to 100 points. A score of 0 indicates that dizziness has no impact on daily life, while a score of 100 signifies a significant impact. The DHI has demonstrated strong psychometric properties, including high test-retest reliability (intrarater correlation coefficient [ICC] 0.72-0.97) and internal consistency reliability (α = 0.72-0.89) (Jacobson & Newman, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Lytras, PhD, Principal Investigator — International Hellenic University
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic Universit, Thessaloniki, Sindos Thessaloníki, Greece, Greece

IPD SHARING:
Plan to Share IPD: No